CLINICAL TRIAL: NCT00268853
Title: Cyclophosphamide, Doxorubicin, Vincristine, Prednisone Plus Rituximab (CHOP-R) and Cyclophosphamide, Pixantrone, Vincristine, Prednisone Plus Rituximab (CPOP-R) in Patients With Diffuse Large-B-cell Lymphoma: A Phase II, Randomized, Multicenter, Comparative Trial
Brief Title: A Trial in Patients With Diffuse Large-B-cell Lymphoma Comparing Pixantrone Against Doxorubicin
Acronym: RAPID
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: CTI BioPharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PIX203
Record Dates: First submitted 2005-12-21; First posted 2005-12-23 (Estimated); Results first posted 2024-05-30 (Actual); Last update posted 2024-05-30 (Actual); Status verified 2024-05

CONDITIONS: Diffuse Large-Cell Lymphoma
Keywords: lymphoma; NHL; large cell; phase II; CHOP R; CPOP R; non Hodgkins
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse; Lymphoma | interventions — R-CHOP protocol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental)
  Interventions: Drug: CPOP-R
- 2 (Active Comparator)
  Interventions: Drug: CHOP-R

INTERVENTIONS:
Drug: CPOP-R — Cyclophosphamide 750 mg/m2, pixantrone 150 mg/m2, vincristine 1.4 mg/m2, rituximab 375 mg.m2 on Day 1 of a 21 day cycle, for 8 cycles Prednisone 100 mg/day on Day 1-5 of a 21 day cycle for 8 cycles
  Arms: 1
Drug: CHOP-R — Cyclophosphamide 750 mg/m2, doxorubicin 50 mg/m2, vincristine 1.4 mg/m2, rituximab 375 mg.m2 on Day 1 of a 21 day cycle, for 8 cycles Prednisone 100 mg/day on Day 1-5 of a 21 day cycle for 8 cycles
  Arms: 2

SUMMARY:
The purpose of this study is to compare the standard CHOP-R regimen of Cyclophosphamide, Doxorubicin, Vincristine, Prednisone, and Rituximab to CPOP-R (same regimen, but substituting Doxorubicin with Pixantrone). The objective is to show that CPOP-R is not inferior to CHOP-R.

DETAILED DESCRIPTION:
In preclinical studies, pixantrone has shown significantly less cardiotoxicity than other anthracyclines or anthracenediones. In addition, patients with relapsed disease, who have received prior maximum doses of anthracyclines, have tolerated high doses of pixantrone with minimal added cardiotoxicity. Pixantrone is currently being studied in a Phase III study in 3rd line aggressive NHL.

ELIGIBILITY:
Inclusion Criteria:

1. Previously untreated and histologically confirmed diffuse large B-cell lymphoma according to REAL/WHO classification.
2. Stage II, III or IV disease
3. CD20+
4. Age ≥ 18 years
5. ECOG performance status ≤ 2
6. At least one objectively bidimensionally measurable lesion as demonstrated by CT, spiral CT, or MRI that can be followed for response as target lesion. Patients with the following sites of disease are NOT eligible:

   * Patients with only skin lesions or only palpable lymph nodes.
   * Patients with spleen or bone marrow as only site of disease.
7. Life expectancy ≥ 3 months
8. Serum bilirubin ≤ 1.5 x the institution's upper limit normal (ULN) and creatinine ≤ 2.0 ULN and AST or ALT ≤ 2.0 x the institution's ULN. If hepatic involvement by lymphoma is present, AST or ALT may be ≤ 5.0 x the institution's ULN.
9. LVEF ≥ 50% determined by MUGA scan.
10. Ability to comply with the visit schedule and assessments required by the protocol.
11. Signed approved informed consent, with understanding of study procedures.

Exclusion Criteria:

1. Any prior chemotherapy (except intrathecal chemotherapy at diagnosis and pretreatment corticosteroid therapy) or radiotherapy: Patients may receive corticosteroid pretreatment therapy for up to 7 days after randomization, pending Investigator's decision to reduce tumor burden.
2. Histological diagnosis of T-cell lymphoma or any B-cell lymphoma other than diffuse large B-cell.
3. History of indolent lymphoma
4. Active CNS involvement based on clinical evaluation .
5. HIV-related lymphoma.
6. Major thoracic and/or abdominal surgery within the 4 weeks before randomization from which the patient has not fully recovered except for diagnosis of NHL. Patients who have had minor surgery may be enrolled after a ≥ 1 week recovery period except for diagnosis of NHL.
7. Clinically significant cardiovascular abnormalities
8. Serious (NCI CTCAE grade 3-4) intercurrent infection at randomization or deep seated or systemic mycotic infections.
9. Clinical symptoms suggesting unresolved HIV, HBV or HCV infection. Patients with seropositivity presumed to be due to prior vaccination against Hepatitis B virus or resolved infection will not be excluded.
10. Active or history of another malignancy except cured basal cell carcinoma of skin or carcinoma in situ of uterine cervix. Patients who have been in remission from another previous malignancy for >5 years will be considered eligible.
11. Known hypersensitivity to the excipients or the study drugs that the patient will receive.
12. Any contraindications to the study drugs as described in the Summary of Product Characteristics or package inserts. 13. Neurological contraindication to vincristine (e.g. peripheral neuropathy).

14. Any condition which, in the judgment of the Investigator, would place the subject at undue risk, interfere with the results of the study, or make the subject otherwise unsuitable. 15. General status that, in the opinion of the Investigator does not permit the administration of eight courses of CHOP-R/CPOP-R. 16. Treatment with any other investigational study drug within 30 days before randomization. Patient must have recovered from all side effects of other investigational therapy. 17. Potentially fertile men and women and their sexual partners not willing to use adequate contraception as defined by the Investigator during the study and for 6 months after the last day of study drug administration.

18. Any circumstance at the time of study entry that would preclude completion of the study or the required follow-up.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 124 (Actual)
Dates: Start 2005-11; Primary Completion 2012-05 (Actual); Study Completion 2012-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gabor Jurida, M.D., Study Director — CTI BioPharma
Locations (75):
- United States (58):
  - Bay Medical Oncology & Hematology, Concord, California
  - Hazel Hawkins Hospital, Dept. of Medical Oncology, Hollister, California
  - UCSD Moore's Cancer Center-Blood & Marrow Transplantation Division, La Jolla, California
  - Loma Linda University Medical Center, Loma Linda, California
  - Hematology/Oncology Group of Orange County, Orange, California
  - Sharp Memorial Hospital, San Diego, California
  - Rocky Mountain Cancer Center, Denver, Colorado
  - The Center of Hematology and Oncology, Boca Raton, Florida
  - Broward Oncology Associates, Fort Lauderdale, Florida
  - Osceola Cancer Center, Kissimmee, Florida
  - Watson Clinic for Cancer Care and Research, Lakeland, Florida
  - Watson Clinic, Lakeland, Florida
  - Memorial Cancer Institute, Pembroke Pines, Florida
  - Hematology Oncology Associates of the Treasure Coast, Port Saint Lucie, Florida
  - Oncology Hematology Associates of West Broward, Tamarac, Florida
  - Hematology Oncology Specialists, Tampa, Florida
  - John B. Amos Cancer Center, Columbus, Georgia
  - Columbus Clinic, Columbus, Georgia
  - Oncology Hematology of Northern Illinois, Gurnee, Illinois
  - Mid-Illinois Hematology & Oncology Associates, Normal, Illinois
  - Cancer Care Center, New Albany, Indiana
  - Consultants in Blood Disorders and Cancer, Louisville, Kentucky
  - Western Kentucky Hematology/Oncology Group, Paducah, Kentucky
  - Our Lady of the Lake Regional Medial Center, Hematology Oncology, Baton Rouge, Louisiana
  - Greater Baltimore Medical Center, Baltimore, Maryland
  - Maryland Hematology/Oncology Associates, PA, Baltimore, Maryland
  - Center for Cancer and Blood Disorders, P.C., Bethesda, Maryland
  - Frederick Memorial Hospital Cancer Center, Frederick, Maryland
  - Tufts-New England Medical Center-The Neely Ctr for Clinical Cancer Research, Boston, Massachusetts
  - Hubert H Humphrey Cancer Center, Robbinsdale, Minnesota
  - North Missssppi Hematology Oncology Associates, Tupelo, Mississippi
  - Capital Comprehensive Cancer Care, Jefferson City, Missouri
  - Southeast Nebraska Hematology and Oncology Consultants, P.C., Lincoln, Nebraska
  - Nevada Cancer Institute, Las Vegas, Nevada
  - New Mexico Hematology/Oncology Consultants, Albuquerque, New Mexico
  - St. Luke's Roosevelt Hospital, New York, New York
  - Interlake Foundation, Inc., Rochester, New York
  - Jacobi Medical Center Phase I Oncology, The Bronx, New York
  - Our Lady of Mercy Medical Center, The Bronx, New York
  - Duke University Medical Center, Durham, North Carolina
  - Brody School of Medicine at East Carolina University - Leo W. Jenkins Cancer Center, Greenville, North Carolina
  - Cancer Treatment & Research Mid-Dakota Clinic, Bismarck, North Dakota
  - Summa Health Systems Hospitals, Akron, Ohio
  - Barberton Citizen's Hospital, Barberton, Ohio
  - Oncology Partners Network, Cincinnati, Ohio
  - Dayton Clinical Oncology Program, Dayton, Ohio
  - Northwest Kaiser Permanente, Portland, Oregon
  - Berks Hematology-Oncology Associates Ltd., Reading, Pennsylvania
  - Charleston Cancer Center, Charleston, South Carolina
  - Low County Hematology & Oncology, Mt. Pleasant, South Carolina
  - The Family Cancer Center, Collierville, Tennessee
  - Thompson Cancer Survival Center, Knoxville, Tennessee
  - Sarah Cannon Cancer Center, Nashville, Tennessee
  - Southwest Regional Cancer Center, Austin, Texas
  - Texas Hematology Oncology Center, Dallas, Texas
  - The Center for Cancer and Blood Disorders, Fort Worth, Texas
  - Northern Utah Hematology Oncology, P.C., Ogden, Utah
  - Multicare Oncology Hematology Specialists, Tacoma, Washington
- Canada (3):
  - London Health Science Center Regional Care Program, London, Ontario
  - The Ottawa Hospital, Ottawa, Ontario
  - Queen Elizabeth II HSC, Halifax
- France (2):
  - CHU Hotel Dieu, Nantes
  - Hopitaux Universitaires de Strabourg - Hopital Hautepierre, Strasbourg
- Germany (5):
  - Klinikum der Universitaet zu Koeln, Cologne
  - Universitaetsklinikum Carl Gustav Carus, Dresden
  - Universitaetsklinikum Duesseldorf, Düsseldorf
  - Klinikum Nurnberg Nord - Medizinische, Nuremberg
  - Universitaetsklinikum Wuerzburg, Würzburg
- Italy (7):
  - Instituto di Ematologia "Lorenzo e Ariosto", Bologna
  - Azienda Ospedaliera Careggi, Florence
  - Farmacia Osepdaliera, Odpedale Umberto I, Mestre
  - Ospedal V. Cervello, Palermo
  - Uiversita La Sapienza, Roma
  - Policlinico S. Maria alle Scotte, Siena
  - Ospedale Civile, Udine

REFERENCES:
- [Result] Herbrecht R, Cernohous P, Engert A, Le Gouill S, Macdonald D, Machida C, Myint H, Saleh A, Singer J, Wilhelm M, van der Jagt R. Comparison of pixantrone-based regimen (CPOP-R) with doxorubicin-based therapy (CHOP-R) for treatment of diffuse large B-cell lymphoma. Ann Oncol. 2013 Oct;24(10):2618-2623. doi: 10.1093/annonc/mdt289. Epub 2013 Aug 14. PMID 23946328

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | CPOP-R | CHOP-R
Started | 61 | 63
Completed | 45 | 44
Not Completed | 16 | 19

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | CPOP-R | CHOP-R | Total
Number analyzed (Participants) | 61 | 63 | 124
Age, Customized [Count of Participants; unit: Participants]
  ≤ 65 Years | 26 | 29 | 55
  >65 Years | 35 | 34 | 69
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 29 | 34 | 63
  Male | 32 | 29 | 61
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Caucasian | 51 | 58 | 109
  Hispanic | 6 | 2 | 8
  Black | 2 | 0 | 2
  Asian | 1 | 0 | 1
  Other | 1 | 3 | 4

OUTCOME MEASURES:

1. Primary Outcome: Response Rate
Time Frame: Subjects followed for 5 years post treatment
Population: Intent to Treat Population
Measure: Count of Participants; unit: Participants
Arm/Group | CPOP-R | CHOP-R
Number analyzed (Participants) | 61 | 63
Participants
  Complete Response | 24 | 28
  Complete Response Unconfirmed | 20 | 22
  Response Rate | 44 | 50

2. Secondary Outcome: Overall Survival
Description: Overall Survival time frame is from the interval between the date of randomization and death due to any cause and measures the total number of deaths.
Time Frame: The interval between the date of randomization and death due to any cause (up to 100 weeks)
Population: Intent to Treat (ITT) Population
Measure: Count of Participants; unit: Participants
Arm/Group | CPOP-R | CHOP-R
Number analyzed (Participants) | 61 | 63
Participants | 18 | 9

3. Secondary Outcome: Median Progression Free Survival (PFS)
Description: The interval between the date of randomization and the event of disease progression or relapse, institution of a new anticancer treatment or death.
Time Frame: From the date of randomization to the first documented disease progression or death (up to 100 weeks)
Population: Intent to Treat Population
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | CPOP-R | CHOP-R
Number analyzed (Participants) | 61 | 63
months | NA [8.6 to NA] — The median survival time is defined to be the time at which the survival curve crosses 50% survival. The curve did not cross 50% (because survival is greater than 50% at the last time point), then median survival is simply non-estimable.The upper CI is non-estimable because there are not sufficient patients contributing events to estimate the upper bound of the confidence interval. | 17.3 [13.3 to NA] — The upper CI is non-estimable because there are not sufficient patients contributing events to estimate the upper bound of the confidence interval.

4. Secondary Outcome: Overall Objective Response Rate
Time Frame: Subjects followed for 5 years post treatment
Population: Intent to Treat Population
Measure: Count of Participants; unit: Participants
Arm/Group | CPOP-R | CHOP-R
Number analyzed (Participants) | 61 | 63
Participants | 50 | 55

5. Secondary Outcome: Time to Treatment Failure
Time Frame: Subjects followed for 5 years post treatment
Population: Intent to Treat Population
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | CPOP-R | CHOP-R
Number analyzed (Participants) | 61 | 63
Months | 30.3 [7.7 to NA] — The upper CI is not estimable because there are not sufficient patients contributing events to estimate the upper bound of the confidence interval | 40.1 [15.1 to NA] — The upper CI is not estimable because there are not sufficient patients contributing events to estimate the upper bound of the confidence interval

ADVERSE EVENTS:
Description: Safety Population
Arm/Group | CPOP-R | CHOP-R
All-Cause Mortality (participants affected / at risk) | 18/59 | 9/63
Serious Adverse Events (participants affected / at risk) | 28/59 | 26/63
Other Adverse Events (participants affected / at risk) | 59/59 | 63/63
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CPOP-R (N=59) | CHOP-R (N=63)
Pneumonia (Infections and infestations) | 4 (4) | 2 (2)
Sepsis (Infections and infestations) | 3 (3) | 1 (1)
Pyelonephritis (Infections and infestations) | 0 (0) | 2 (2)
Urinary Tract Infection (Infections and infestations) | 1 (1) | 1 (1)
Bacterial Sepsis (Infections and infestations) | 0 (0) | 1 (1)
Bronchitis (Infections and infestations) | 1 (1) | 0 (0)
Cellulitis (Infections and infestations) | 1 (1) | 0 (0)
Clostridial Infection (Infections and infestations) | 1 (1) | 0 (0)
Escherichia Sepsis (Infections and infestations) | 0 (0) | 1 (1)
Infection (Infections and infestations) | 1 (1) | 0 (0)
Oesophageal Candidiasis (Infections and infestations) | 1 (1) | 0 (0)
Otitis Externa (Infections and infestations) | 0 (0) | 1 (1)
Psoas Abscess (Infections and infestations) | 0 (0) | 1 (1)
Thrombophlebitis Septic (Infections and infestations) | 1 (1) | 0 (0)
Urosepsis (Infections and infestations) | 0 (0) | 1 (1)
Wound Infection (Infections and infestations) | 1 (1) | 0 (0)
Oncocytoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 8 (8) | 9 (9)
Febrile Neutropenia (Blood and lymphatic system disorders) | 7 (7) | 8 (8)
Anaemia (Blood and lymphatic system disorders) | 3 (3) | 2 (2)
Leukopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 2 (2) | 2 (2)
Hypoglycaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Type 2 Diabetes Mellitus (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Anxiety (Psychiatric disorders) | 1 (1) | 0 (0)
Depression (Psychiatric disorders) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 2 (2) | 0 (0)
Amyotrophic Lateral Sclerosis (Nervous system disorders) | 1 (1) | 0 (0)
Cerebral Ischemia (Nervous system disorders) | 1 (1) | 0 (0)
Convulsion (Nervous system disorders) | 1 (1) | 0 (0)
Presyncope (Nervous system disorders) | 1 (1) | 0 (0)
Somnolence (Nervous system disorders) | 1 (1) | 0 (0)
Transient Ischaemic Attack (Nervous system disorders) | 1 (1) | 0 (0)
Cardiac Arrest (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac Failure Congestive (Cardiac disorders) | 0 (0) | 1 (1)
Deep Vein Thrombosis (Vascular disorders) | 1 (1) | 4 (4)
Thrombophlebitis (Vascular disorders) | 0 (0) | 2 (2)
Lymphoedema (Vascular disorders) | 1 (1) | 0 (0)
Orthostatic Hypotension (Vascular disorders) | 0 (0) | 1 (1)
Thrombophlebitis Superficial (Vascular disorders) | 1 (1) | 0 (0)
Thrombosis (Vascular disorders) | 0 (0) | 1 (1)
Vena Cava Thrombosis (Vascular disorders) | 0 (0) | 1 (1)
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 3 (3)
Acute Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Lung Disorder (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pulmonary Oedema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastrointestinal Haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Oesophagitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Peritoneal Effusion (Gastrointestinal disorders) | 0 (0) | 1 (1)
Small Intestinal Perforation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0)
Back Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Bone Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Urinary Bladder Haemorrhage (Renal and urinary disorders) | 1 (1) | 0 (0)
Urinoma (Renal and urinary disorders) | 0 (0) | 1 (1)
Prostatitis (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Familial Mediterranean Fever (Congenital, familial and genetic disorders) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 3 (3) | 5 (5)
Asthenia (General disorders) | 1 (1) | 0 (0)
Mucosal Inflammation (General disorders) | 0 (0) | 1 (1)
Non-cardiac Chest Pain (General disorders) | 1 (1) | 0 (0)
Ejection Fraction Decreased (Investigations) | 1 (1) | 1 (1)
Liver Function Test Abnormal (Investigations) | 0 (0) | 1 (1)
Neutrophil Count Decreased (Investigations) | 1 (1) | 0 (0)
Platelet Count Decreased (Investigations) | 1 (1) | 0 (0)
White Blood Cell Count Decreased (Investigations) | 1 (1) | 0 (0)
Clavicle Fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Facial Bones Fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CPOP-R (N=59) | CHOP-R (N=63)
Urinary Tract Infection (Infections and infestations) | 5 (5) | 4 (4)
Bronchitis (Infections and infestations) | 3 (3) | 3 (3)
Candidiasis (Infections and infestations) | 3 (3) | 4 (4)
Nasopharyngitis (Infections and infestations) | 4 (4) | 3 (3)
Rhinitis (Infections and infestations) | 3 (3) | 3 (3)
Oral Candidiasis (Infections and infestations) | 0 (0) | 4 (4)
Neutropenia (Blood and lymphatic system disorders) | 30 (30) | 33 (33)
Anaemia (Blood and lymphatic system disorders) | 23 (23) | 20 (20)
Leukopenia (Blood and lymphatic system disorders) | 17 (17) | 16 (16)
Thrombocytopenia (Blood and lymphatic system disorders) | 8 (8) | 13 (13)
Lymphopenia (Blood and lymphatic system disorders) | 10 (10) | 8 (8)
Hypokalaemia (Metabolism and nutrition disorders) | 12 (12) | 10 (10)
Anorexia (Metabolism and nutrition disorders) | 12 (12) | 11 (11)
Dehydration (Metabolism and nutrition disorders) | 8 (8) | 8 (8)
Hyperglycaemia (Metabolism and nutrition disorders) | 7 (7) | 6 (6)
Decreased Appetite (Metabolism and nutrition disorders) | 5 (5) | 1 (1)
Hypocalcaemia (Metabolism and nutrition disorders) | 3 (3) | 3 (3)
Hyperuricaemia (Metabolism and nutrition disorders) | 4 (4) | 1 (1)
Hyponatraemia (Metabolism and nutrition disorders) | 3 (3) | 2 (2)
Insomnia (Psychiatric disorders) | 6 (6) | 13 (13)
Anxiety (Psychiatric disorders) | 3 (3) | 3 (3)
Depression (Psychiatric disorders) | 3 (3) | 2 (2)
Headache (Nervous system disorders) | 13 (13) | 14 (14)
Paraesthesia (Nervous system disorders) | 9 (9) | 12 (12)
Neuropathy Peripheral (Nervous system disorders) | 13 (13) | 6 (6)
Dizziness (Nervous system disorders) | 8 (8) | 8 (8)
Dysgeusia (Nervous system disorders) | 6 (6) | 7 (7)
Peripheral Sensory Neuropathy (Nervous system disorders) | 6 (6) | 4 (4)
Hypoaesthesia (Nervous system disorders) | 6 (6) | 3 (3)
Hyporeflexia (Nervous system disorders) | 5 (5) | 4 (4)
Polyneuropathy (Nervous system disorders) | 5 (5) | 3 (3)
Conjunctivitis (Eye disorders) | 3 (3) | 1 (1)
Hypertension (Vascular disorders) | 3 (3) | 5 (5)
Cough (Respiratory, thoracic and mediastinal disorders) | 8 (8) | 14 (14)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 9 (9)
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 4 (4)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 4 (4)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 0 (0)
Nausea (Gastrointestinal disorders) | 24 (24) | 23 (23)
Constipation (Gastrointestinal disorders) | 18 (18) | 20 (20)
Vomiting (Gastrointestinal disorders) | 10 (10) | 15 (15)
Diarrhoea (Gastrointestinal disorders) | 10 (10) | 12 (12)
Abdominal Pain (Gastrointestinal disorders) | 8 (8) | 7 (7)
Dyspepsia (Gastrointestinal disorders) | 7 (7) | 8 (8)
Stomatitis (Gastrointestinal disorders) | 4 (4) | 11 (11)
Abdominal Pain Upper (Gastrointestinal disorders) | 4 (4) | 4 (4)
Dysphagia (Gastrointestinal disorders) | 3 (3) | 4 (4)
Gastritis (Gastrointestinal disorders) | 2 (2) | 4 (4)
Bone Pain (Musculoskeletal and connective tissue disorders) | 11 (11) | 7 (7)
Back Pain (Musculoskeletal and connective tissue disorders) | 10 (10) | 4 (4)
Alopecia (Skin and subcutaneous tissue disorders) | 26 (26) | 25 (25)
Skin Discolouration (Skin and subcutaneous tissue disorders) | 14 (14) | 0 (0)
Night Sweats (Skin and subcutaneous tissue disorders) | 3 (3) | 4 (4)
Rash (Skin and subcutaneous tissue disorders) | 3 (3) | 4 (4)
Nail Disorder (Skin and subcutaneous tissue disorders) | 3 (3) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 8 (8) | 6 (6)
Muscular Weakness (Musculoskeletal and connective tissue disorders) | 6 (6) | 6 (6)
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 5 (5) | 5 (5)
Muscle Spasms (Musculoskeletal and connective tissue disorders) | 4 (4) | 4 (4)
Myalgia (Musculoskeletal and connective tissue disorders) | 4 (4) | 4 (4)
Pain in Jaw (Musculoskeletal and connective tissue disorders) | 3 (3) | 1 (1)
Musculoskeletal Pain (Musculoskeletal and connective tissue disorders) | 3 (3) | 0 (0)
Pollakiuria (Renal and urinary disorders) | 1 (1) | 8 (8)
Chromaturia (Renal and urinary disorders) | 7 (7) | 0 (0)
Pyrexia (General disorders) | 11 (11) | 12 (12)
Asthenia (General disorders) | 18 (18) | 16 (16)
Mucosal Inflammation (General disorders) | 3 (3) | 6 (6)
Fatigue (General disorders) | 26 (26) | 25 (25)
Oedema Peripheral (General disorders) | 12 (12) | 12 (12)
Chest Pain (General disorders) | 2 (2) | 4 (4)
Chills (General disorders) | 2 (2) | 4 (4)
Influenza-like Illness (General disorders) | 3 (3) | 3 (3)
Ejection Fraction Decreased (Investigations) | 18 (18) | 19 (19)
Weight Decreased (Investigations) | 11 (11) | 7 (7)
Alanine Aminotransferase Increased (Investigations) | 3 (3) | 2 (2)
Aspartate Aminotransferase Increased (Investigations) | 3 (3) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No